CLINICAL TRIAL: NCT06797648
Title: Epidemiology of Infection in AML, A European Haematology Association Survey
Brief Title: Epidemiology of Infection in Acute Myeloid Leukemia (AML)
Acronym: EPIAMLINF
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7283
Record Dates: First submitted 2025-01-23; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data analysis — follow up after 15 months

SUMMARY:
In recent years, multiple factors have strongly impacted the epidemiology of infections in patients with acute myeloid leukemia. On the one hand, the availability of new effective antileukemic drugs (i.e. venetoclax, FLT-3 inhibitors, CPX-351) have expanded the pharmacological armamentarium. On the other hand, first, many of them inhere drug-drug interactions with azoles and fluoroquinolones, facing clinicians with the choice of whether to administer antimicrobial prophylaxis or not. Secondly, there is an increase in infections due to multi-resistant agents from both the bacterial and fungal field. Third, the onset of a viral pandemic that had high relevance in these patients in terms of morbidity and mortality.

The aim of this survey is to collect information on the largest possible sample of patients with AML during induction/consolidation/relapsed-refractory treatment, regarding bacterial, viral, fungal infections. We will evaluate the incidence of the various types of infection in relation to the type of treatment that patients will undergo, in order to identify what should be the best antimicrobial prophylactic approach in each subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to sign the consent form
* Age ≥18 years
* New diagnosis of AML (only cases diagnosed after 01/03/2025), APL are included
* Patients not elegible to any kind of chemotherapy but only best supportive care (BSC)
* AML patients treated with induction treatment, consolidation treatment, or relapsed/refractory (for these latter patients the first diagnosis must not be prior to March 01, 2025)
* All kind of infectious diseases, including parasites.
* Clincally or microbiologically diagnosed infections, including FUO

Exclusion Criteria:

* Hematological diseases, other than AML
* Patients with an AML diagnosis prior to March 2025 but who relapsed during the period under examination
* Patients relapsed after allo or auto-HSCT (Inclusion of post-transplant patients would create an evaluation bias due to the immunological alterations that the transplant procedure causes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population must be ≥18 years of age with a new diagnosis AML and microbiologically/clinically documented bacterial/fungal/viral infection. Patients with fever of unidentified origin (FUO) could be included. In order to obtain a denominator for all cases of AML, it is required to fill out the eCRF. The form must be filled out for each phase of treatment (i.e. induction, consolidation, relapsed, refractory). Patients stop recording when they go to HSCT.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of bacterial/fungal/viral infections in AML patients | 18 months
  To evaluate the incidence of bacterial/fungal/viral infections in AML patients undergoing induction, consolidation or salvage chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: LIVIO PAGANO, PROF, Principal Investigator — FONDAZIONE POLICLINICO GEMELLI, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli Irccs, Uoc Ematologia, Rome, Italy